CLINICAL TRIAL: NCT07336225
Title: Prognostic Value of Cardiovascular Magnetic Resonance in Patients With Cardiac Implantable Electronic Devices
Brief Title: CMR-Based Prognostic Study in Patients With Cardiac Implantable Electronic Devices
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-CIED
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Implantable Electronic Device Cohort
  Interventions: Other: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging — Cardiac magnetic resonance imaging performed as part of routine clinical care. Imaging data are used for observational research analyses only, without altering clinical management.

SUMMARY:
Cardiac implantable electronic devices (CIEDs) are widely used to treat patients with heart failure, malignant arrhythmias, and other conditions. However, accurately identifying suitable candidates for CIED implantation remains a clinical challenge. Cardiovascular magnetic resonance imaging (CMR) provides a comprehensive assessment of cardiac structure, function, and tissue characteristics, facilitating evaluation of the myocardial substrate for arrhythmias. This study aims to evaluate the prognostic value of multiparametric CMR-derived imaging markers in CIED patients through preoperative CMR examinations. Imaging parameters of interest include structural-functional indices, myocardial strain, late gadolinium enhancement, entropy, and T1 and T2 mapping. Long-term clinical outcomes will be obtained from existing medical records and follow-up. The primary endpoint is sudden cardiac death (SCD) or SCD-equivalent events, defined as SCD, resuscitated cardiac arrest, sustained ventricular tachycardia or ventricular fibrillation, or appropriate ICD therapy. Secondary endpoints include all-cause mortality or heart failure rehospitalization. This study aims to elucidate the role of CMR in assessing CIED treatment indications and long-term risk stratification, thereby helping to optimize CIED implantation decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old).
2. Patients with guideline-based indications for cardiac implantable electronic device (CIED) therapy, including pacemaker, implantable cardioverter-defibrillator, or cardiac resynchronization therapy.
3. Patients who underwent cardiovascular magnetic resonance (CMR) imaging as part of routine clinical evaluation prior to CIED implantation or consideration of CIED therapy.

Exclusion Criteria:

1. Patients younger than 18 years of age.
2. Patients with non-diagnostic or poor-quality CMR images that preclude reliable image analysis.
3. Patients with incomplete key clinical data or missing follow-up information for primary outcome assessment.
4. Patients with prior heart transplantation or implantation of ventricular assist devices before CMR examination.
5. Patients with congenital heart disease requiring surgical correction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population includes patients meeting indications for cardiac implantable electronic devices (CIEDs), encompassing those with indications for pacemakers, implantable cardioverter defibrillators, or cardiac resynchronization therapy. This cohort will include individuals with multiple underlying conditions such as heart failure, arrhythmias, or conduction disorders like left bundle branch block, which clinically necessitate the implantation of CIEDs.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of sudden cardiac death (SCD) and SCD-equivalent events | 1-10 years
  SCD, defined as unexpected death within ≤1 hour of cardiac symptoms in the absence of any progressive cardiac deterioration, during sleep, or ≤24 hours of last being seen alive. SCD-equivalent events, defined as an appropriate implantable cardioverter defibrillator shock for ventricular arrhythmia, a nonfatal episode of ventricular fibrillation or spontaneous sustained ventricular tachycardia causing hemodynamic compromise and requiring cardioversion

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, China